CLINICAL TRIAL: NCT04998838
Title: Stop Hep B @ Birth: Community-Oriented Care Model for the Prevention of Mother-To-Child Transmission of Hepatitis B in Peri-Urban Yangon
Brief Title: Stop Hep B @ Birth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Myanmar Liver Foundation (Other)
Responsible Party: Principal Investigator, Khin Pyone Kyi, President, Myanmar Liver Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HBV2020
Record Dates: First submitted 2021-01-19; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; hepatitis B hyperimmune globulin

STUDY DESIGN:
Intervention Model Description: Antenatal screening for HBV, anti-viral treatment with tenofovir according to treatment eligibility criteria, and birth dose vaccination at delivery to prevent mother-to-child transmission of HBV
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tenofovir Disoproxil Fumerate (Experimental): Pregnant women (>=20 weeks of gestation) will be treated with TDF if clinically eligible; newborns will receive birth dose vaccine (and HBIG if eligible). Non-eligible women will be treated according to normal practices; newborns will still receive birth dose vaccine.
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 mg daily; HBV birth dose vaccine; hepatitis B immune globulin (HBIG); Drug: Regular Myanmar treatment

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate 300 mg daily; HBV birth dose vaccine; hepatitis B immune globulin (HBIG) — Antenatal screening for HBV, anti-viral treatment with tenofovir according to treatment eligibility criteria, and birth dose vaccination at delivery to prevent mother-to-child transmission of HBV
  Other Names: Viread
Drug: Regular Myanmar treatment — Treated according to normal Myanmar processes for HBV positive patients

SUMMARY:
Single arm, prospective open-label study of a care model consisting of two components: Component I aims to achieve high coverage of interventions to prevent maternal-to-child transmission of hepatitis B virus: antenatal tenofovir, and timely newborn administration of hepatitis B birth dose vaccine and hepatitis B immune globulin; Component II aims to achieve high coverage of screening, vaccination, and anti-viral therapy for HBV among household members of women with chronic HBV infection.

DETAILED DESCRIPTION:
An estimated 248 million people worldwide are chronically infected with hepatitis B virus (HBV); and 75% of them live in Asia. Mother-to-child transmission (MTCT) accounts for the majority of chronic hepatitis B infections in Southeast Asia. Elimination of MTCT of HBV is theoretically possible with a comprehensive suite of interventions that includes birth dose vaccination, hepatitis B immune globulin, and antenatal antiviral therapy (e.g., tenofovir). However, the ideal gestational age to initiate antenatal tenofovir remains undefined; and evidence is lacking for implementation strategies capable of providing cost-effective, equitable access to a comprehensive suite of interventions to prevent MTCT of HBV in low-resource settings.

Component I: Prevention of Vertical Transmission Pregnant women living in the study area will be identified and screened for hepatitis B by a network of antenatal care (ANC) providers and existing community outreach workers; HBsAg positive patients will be invited to participate in the study. Consenting participants will provide serum samples to assess eligibility for anti-viral therapy: creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), platelet count, HCV, HIV. Pregnant women eligible for antiviral therapy according to WHO criteria, or who have viral load (VL) >200,000 IU/mL, will be treated with tenofovir starting at 20 weeks gestation through 4 weeks postpartum. Hospital-based delivery will be encouraged. All newborns, including those delivered at home, will receive the HBV birth dose vaccine within 24 hours of delivery, and newborns of women on tenofovir treatment will also receive Hepatitis B Immunoglobulin within 24 hours after delivery. Children will be linked to routine immunization services in Myanmar to complete their HBV vaccination series (HBV is co-formulated in a pentavalent vaccine). Maternal VL will be measured at delivery; infants will be tested for hepatitis B infection at 24-28 weeks postpartum.

Component II -- Household Screening and Treatment The household members of HBsAg positive pregnant women who consent to participate in the study will be screened for HBV-related immune status and chronic HBV infection. Non-immune individuals (HBsAb/Ag negative) will be vaccinated; HBsAg positive household members will be assessed for treatment eligibility and initiated on anti-viral therapy according to World Helath Organization guidelines. Eligible household members will also be screened every six months for hepatocellular carcinoma (HCC) by liver ulatrasound and alpha-fetoprotein levels

Qualitative Study:

In-depth interviews with approximately 30 HBsAg-positive women, 30 HBVsAg-negative women, and 20 household members of study participants will be conducted to assess barriers and facilitators related to HBV testing and treatment. Approximately 15 key-informant interviews with healthcare providers and community leaders will also be conducted. Sample size will depend on data saturation and will be adjusted based on results of data analysis during the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women >= 18 years of age
* Gestational age =<34 weeks
* Test positive for HBsAg
* Live in study site area in South Dagon and Dagon Seikkan Townships, Yangon Region
* Give informed consent to participate in the study
* Newborns and household members of pregnant women enrolled in the study according to previous inclusion criteria

Exclusion Criteria:

* Alanine aminotransferase (ALT) levels >300 IU/L

For qualitative study:

Inclusion criteria

* Key informants (e.g., healthcare providers and community leaders in the study area) OR
* HBsAg+ women and their household members in the study area
* HBsAg- women and their household members in the stud area
* Give informed consent to participate in the study
* History of renal dysfunction
* CrCL < 50mL/min
* ALT>5 times the upper limit of normal (ULN)
* Evidence of decompensated cirrhosis (e.g., jaundice, ascites, history of upper gastrointestinal bleeding/esophageal varices, and hepatic encephalopathy)
* Any concomitant condition or treatment that, in view of the clinical site investigator, would contraindicate participation or satisfactory follow-up in the study HIV positive status unless 1) they are currently on additional ART therapy, or 2) their viral load is demonstrated to be <50 copies. Women who are newly diagnosed with HIV and referred to start a TDF-based regimen may be considered eligible once they have started the TDF-based regimen.
* Concurrent participation in any other clinical trial without written agreement of the study team
* Does not intend to deliver within catchment area, and/or intends to migrate before newborn follow-up is complete

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Vaccine within 24 hours | Within 24 hours of birth
  Proportion of newborns of HBsAg positive mothers receiving HBV vaccine within 24 hours of birth
Effective treatment of pregnant women | During pregnancy (until delivery) of each woman, average of 9 months
  Proportions of pregnant women with chronic HBV (HBsAg positive) who are (a) linked to care (attend BK Kee Clinic for assessment of treatment eligibility); (b) complete TDF eligibility testing; (c) initiate tenofovir treatment (TDF, among those eligible); (d) adhere to TDF treatment until delivery and (e) continue treatment until 4 weeks post-partum
  o Low/medium/high high medication adherence are defined, respectively, as ≤6, 6-7 or 8 points on the Morisky Medication Adherence Scale (MMAS-8)
Household contact screening | Upon identification of participating women, until the end of the project, average of 1 year
  Proportions of adult household contacts who (a) are screened for chronic HBV infection and immunity (HBsAg/Ab); (b) are linked to care (among HBsAg positive) or vaccinated (if HBsAb negative); (c) complete appropriate testing for hepatocellular carcinoma (HCC) screening, (d) eligible for TDF treatment; (e) initiate chronic HBV treatment with TDF

SECONDARY OUTCOMES:
Total screening of mothers | During pregnancy (until delivery) of each woman, average of 9 months
  Proportion of pregnant women in the target population who are:
  * screened for HBsAg (denominator estimated from population census counts and crude birth rate)
  * HBsAg positive (chronic HBV prevalence among women attending ANC)
Antenatal care for HBV positive pregnant mothers | During pregnancy (until delivery) of each woman, average of 9 months
  Proportions of pregnant women with chronic HBV who:
  * attend their first antenatal care (ANC) visit prior to 20, 24, 28 and 32 weeks gestation
  * are eligible for TDF (HBV VL >200,00 IU/mL or WHO criteria)
  * are HBeAg positive
  * deliver at home
Vaccination of HBV negative pregnant mothers | During pregnancy (until delivery) of each woman, average of 9 months
  Proportion of women who tested negative for HBsAg and HBsAb at baseline who complete the HBV vaccination schedule
Treatment of high viral load pregnant mothers | At delivery; during antenatal care testing; at 4 months postpartum, throughout the project, average of 12 months
  Among women who had VL>200,000 IU/mL at baseline and were eligible for TDF treatment:
  * the proportion that achieve viral suppression (HBV DNA <200,000 IU/mL) at delivery
  * the proportion who are HBeAg positive
  * proportion with HBV flare 4 months postpartum (ALT >300 IU/L)
Viral suppression | At delivery, throughout the project (one off)
  Associations of maternal viral suppression (VL <200,000 at delivery and: baseline HBV VL, duration of exposure to TDF, and TDF adherence
Mother-to-child transmission | At 28 weeks postpartum, throughout the project (one off)
  Proportion of infants born to HBsAg positive mothers who
  * complete the HBV vaccination series within the recommended intervals
  * are HBsAg positive or with measurable HBV VL at 28 weeks postpartum (rate of mother-to-child transmission of HBV)
Household screening | At household screening, throughout the project (one off)
  Among household members screened for HBsAg and HBsAb:
  o Prevalence of chronic infection (% HBsAg positive); and immune status (% HBsAb positive and HBsAg negative)

OTHER OUTCOMES:
Completed vaccination courses | Before age 1, average of 1 year
  Proportion of infants of HBsAg positive mothers who complete HBV vaccination prior to study termination, before and after coronavirus- and coup- related delays in public vaccination program
Proportion of pregnant women with HBsAg identified by surveillance team members | During pregnancy, average of 9 months
  Proportion of pregnant women with HBsAg identified by surveillance team members
Timeliness of pregnancy surveillance | During pregnancy, average of 9 months
  Among pregnant women identified by surveillance team members:
  * Proportion who are linked to care and screened for HBsAg
  * Proportions identified prior to gestational age of 20, 24, 28 and 32 weeks
Equity of intervention | During pregnancy and in first year after delivery, average of 16 months
  Distributions of select outcomes according to age, sex and axes of social disadvantage: household wealth; educational attainment; occupation; and ethnic/religious affiliation

CONTACTS AND LOCATIONS:
Overall Officials: Khin Phone Kyi, MD, Principal Investigator — Myanmar Liver Foundation; Adam K Richards, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- BK Kee Clinic, Yangon, Burma

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are currently developing an individual participant data (IPD) sharing plan.